CLINICAL TRIAL: NCT04784429
Title: Assessing Outcomes With Microprocessor Knee Utilization in a K2 Population
Acronym: ASCENT K2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Otto Bock Healthcare Products GmbH (Industry)
Collaborators: Hanger Clinic: Prosthetics & Orthotics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OB113
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Lower Limb Amputation Above Knee (Injury); Congenital Amputation of Lower Limb; Lower Limb Amputation Knee
Keywords: Prosthetic knee, lower limb amputation, microprocessor controlled knee, K2
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MPK (Experimental): Microprocessor controlled knee
  Interventions: Device: Kenevo or C-Leg 4
- NMPK (Active Comparator): Non-microprocessor controlled knee
  Interventions: Device: Non microprocessor controlled knee (NMPK)

INTERVENTIONS:
Device: Kenevo or C-Leg 4 — Kenevo fitted to subjects walking slower than 0.8 m/s as measured by the 2-minute Walk Test. C-Leg 4 fitted to subjects walking faster than 0.8 m/s.
  Arms: MPK
Device: Non microprocessor controlled knee (NMPK) — NMPK consistent with current standards of care
  Arms: NMPK

SUMMARY:
Two-phased randomized controlled trial comparing the impact of microprocessor controlled knee prostheses (MPK) with the impact of non-microprocessor controlled knee prostheses (NPMK) in patients with a transfemoral/knee disarticulation level amputation categorized as K2 ambulators.

DETAILED DESCRIPTION:
Randomized controlled trial investigating the benefits of microprocessor controlled knee prostheses (MPK) in patients with a transfemoral or knee disarticulation level amputation categorized by Medicare Functional Classification Level (MFCL) as a Limited Community Ambulator (K-Level 2). There are two aims for the study. Aim 1 is to understand the effect of MPK technology for the K2 ambulator on reducing fear and anxiety of falling, improving health-related quality of life, and participation in society and activities. Aim 2 is to understand the long-term effect of MPK technology the aspects from Aim 1 as well as reducing morbidity. The trial will be conducted in two phases. Phase 1 will cover the initial 12-month period to address Aim 1, and phase 2 will monitor from 12 months to 5 years to address Aim 2.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transfemoral or knee disarticulation amputation
* Received prosthesis between 4 - 24 months prior
* Currently uses prosthesis
* K2 ambulator status
* Able to speak English or Spanish language
* Age ≥ 65 years at Baseline Assessment (one month after enrollment)
* Minimum Socket Comfort Score (SCS) of 6/10

Exclusion Criteria:

* Upper limb involvement
* Individuals ≥ 275 lbs
* Unable to provide informed consent
* History of acute or chronic residual limb breakdown
* History of 2 or more socket adjustments or replacements in the past 6 months
* Amputation of the contralateral limb
* Active malignancy
* Rapidly declining health status resulting in reduced activity in the past 6 months, as determined by patient's clinician and confirmed by Clinical & Scientific Affairs personnel
* Patient unable or unwilling to follow study procedures
* Pregnant women, institutionalized persons, and children

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 107 (Actual)
Dates: Start 2021-06-11 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Fear of Falling Avoidance Behavior Questionnaire (FFABQ) | 12 months
  This is a 14 item survey assessment originally developed with community-dwelling older adults which measures the degree to which respondents avoid activities due to their fear of falling. Responses are on a 5-point scale with 0 = completely disagree and 4 = completely agree. The total possible score is 56 points. A higher score indicates a greater activity limitation and participation restriction as a result of the fear of falling.
Fear of Falling Avoidance Behavior Questionnaire (FFABQ) | 5 years
  This is a 14 item survey assessment originally developed with community-dwelling older adults which measures the degree to which respondents avoid activities due to their fear of falling. Responses are on a 5-point scale with 0 = completely disagree and 4 = completely agree. The total possible score is 56 points. A higher score indicates a greater activity limitation and participation restriction as a result of the fear of falling.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) - 29 | 12 months
  The survey assessment comprises from 7 health domains (physical function, anxiety, depression, fatigue, sleep disturbance, satisfaction with social roles, and pain interference). The combined constructs serve to provide a measure of patient's quality of life. Raw scores are converted to T-scores which standardizes the scores with a mean of 50 and standard deviation of 10. Being above or below the standard deviation could be desirable or undesirable based on the domain being measured. Higher scores means more of the concept being measured (e.g. more fatigue).
Patient-Reported Outcomes Measurement Information System (PROMIS) - Ability to Participate in Social Roles and Activities (APSRA) | 12 months
  Within the PROMIS system, this specific set of question is aimed at assessing the person's ability to perform usual social roles and activities, a construct noted to be of great significance to well-being within the World Health Organization International Classification of Function model. Four of the PROMIS-APSRA questions are included on the PROMIS-29 within the domain of 'satisfaction with social roles'. The addition of four more questions helps with the responsiveness within this specific domain. Thus the additional four questions of the PROMIS-APSRA will be administered to assess the domain of participation and activity.
12-month fall count from bi-weekly fall journal | 12 months
  On a bi-weekly cadence, individuals will be asked to complete the Lower Limb Amputation Fall Survey. This survey was developed for the purpose of documenting number of falls and near-falls over a given period, as well as insight into the causality.
Average daily step counts | 12 months
  Difference in average daily step activity count from 1 week after initial assessment compared to average daily step activity count for 1 week prior to 12-month assessment. Modern activity monitors provide the ability to translate movement from triaxial inertial measurement units into corresponding step activity with great precision.
Fear of Falling Avoidance Behavior Questionnaire (FFABQ) | 3 years
  This is a 14 item survey assessment originally developed with community-dwelling older adults which measures the degree to which respondents avoid activities due to their fear of falling. Responses are on a 5-point scale with 0 = completely disagree and 4 = completely agree. The total possible score is 56 points. A higher score indicates a greater activity limitation and participation restriction as a result of the fear of falling.
Patient-Reported Outcomes Measurement Information System (PROMIS) - 29 | 5 years
  The survey assessment comprises from 7 health domains (physical function, anxiety, depression, fatigue, sleep disturbance, satisfaction with social roles, and pain interference). The combined constructs serve to provide a measure of patient's quality of life. Raw scores are converted to T-scores which standardizes the scores with a mean of 50 and standard deviation of 10. Being above or below the standard deviation could be desirable or undesirable based on the domain being measured. Higher scores means more of the concept being measured (e.g. more fatigue).
Patient-Reported Outcomes Measurement Information System (PROMIS) - Ability to Participate in Social Roles and Activities (APSRA) | 5 years
  Within the PROMIS system, this specific set of question is aimed at assessing the person's ability to perform usual social roles and activities, a construct noted to be of great significance to well-being within the World Health Organization International Classification of Function model. Four of the PROMIS-APSRA questions are included on the PROMIS-29 within the domain of 'satisfaction with social roles'. The addition of four more questions helps with the responsiveness within this specific domain. Thus the additional four questions of the PROMIS-APSRA will be administered to assess the domain of participation and activity.
10-meter Walk Test (10mWT) | 5 years
  The 10mWT is a standardized test of self-selected walking speed in which patients are timed over the middle 6 meters (19.7 feet) of a 10-meter (32.8 feet) flat walkway. The self-selected walking speed is calculated in meters per second and has been discussed as a potential vital sign given its strong relationship with survival. It will serve as a marker of morbidity.
Timed Up and Go (TUG) | 5 years
  The Timed Up-and-Go test is a standard basic mobility test that includes a sit-to-stand, gait initiation, walking, turning, and stand-to-sit. The test measures, in seconds, the time to stand up from an arm chair, walk a distance of 3 meters (approximately 10 feet), turn, walk back to the chair and sit down. It is a measure of function, has been used to assess the risk of falling, and will serve as a marker of morbidity.
Patient-Reported Outcomes Measurement Information System (PROMIS) - 29 | 3 years
  Difference in average daily step activity count from 1 week after initial assessment compared to average daily step activity count for 1 week prior to 5-year assessment. Modern activity monitors provide the ability to translate movement from triaxial inertial measurement units into corresponding step activity with great precision.
Patient-Reported Outcomes Measurement Information System (PROMIS) - Ability to Participate in Social Roles and Activities (APSRA) | 3 years
  Within the PROMIS system, this specific set of question is aimed at assessing the person's ability to perform usual social roles and activities, a construct noted to be of great significance to well-being within the World Health Organization International Classification of Function model. Four of the PROMIS-APSRA questions are included on the PROMIS-29 within the domain of 'satisfaction with social roles'. The addition of four more questions helps with the responsiveness within this specific domain. Thus the additional four questions of the PROMIS-APSRA will be administered to assess the domain of participation and activity.
10-meter Walk Test (10mWT) | 3 years
  The 10mWT is a standardized test of self-selected walking speed in which patients are timed over the middle 6 meters (19.7 feet) of a 10-meter (32.8 feet) flat walkway. The self-selected walking speed is calculated in meters per second and has been discussed as a potential vital sign given its strong relationship with survival. It will serve as a marker of morbidity.
Timed Up and Go (TUG) | 3 years
  The Timed Up-and-Go test is a standard basic mobility test that includes a sit-to-stand, gait initiation, walking, turning, and stand-to-sit. The test measures, in seconds, the time to stand up from an arm chair, walk a distance of 3 meters (approximately 10 feet), turn, walk back to the chair and sit down. It is a measure of function, has been used to assess the risk of falling, and will serve as a marker of morbidity.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kannenberg, MD, PhD, Principal Investigator — Otto Bock Healthcare Products GmbH; Shane Wurdeman, PhD, Principal Investigator — Hanger Clinic: Prosthetics & Orthotics
Locations (90):
- United States (90):
  - Hanger Clinic - 321 Westgate Pkwy, Dothan, Alabama
  - Hanger Clinic - 3501 S Mercy Road, Gilbert, Arizona
  - Hanger Clinic - 3816 N. 7th St., Phoenix, Arizona
  - Hanger Clinic - 4045 E Bell Rd, Phoenix, Arizona
  - Hanger Clinic - 13925 Meeker Blvd, Suite 5, Sun City West, Arizona
  - Hanger Clinic - 4849 Lonetree Way, STE B, Antioch, California
  - Hanger Clinic - 1743 Creekside, Suite #110, Folsom, California
  - Hanger Clinic - California - 1248 32nd St, Sacramento, California
  - Hanger Clinic - 23451 Madison St., Suite 200, Skypark Building 7, Torrance, California
  - Hanger Clinic - 820 S Akers St, Ste 230, Visalia, California
  - Hanger Clinic - 1215 Plumas Street, Suite 1000, Yuba City, California
  - Hanger Clinic - St. Anthony Hospital - Medical Plaza 1, Suite 230, 11750 West 2nd Place, Lakewood, Colorado
  - Hanger Clinic - 1119 Professional Park Drive, Brandon, Florida
  - Hanger Clinic - 1400 Mason Ave. Suite 103, Daytona Beach, Florida
  - Hanger Clinic - 12591 Creekside Lane, Fort Myers, Florida
  - Hanger Clinic - 221 W. Main Street, Inverness, Florida
  - Hanger Clinic - 308 East Oak Street, Kissimmee, Florida
  - Hanger Clinic - 6270 Naples Blvd, Bldg 1, Naples, Florida
  - Hanger Clinic - 824 Creighton Road, Pensacola, Florida
  - Hanger Clinic - 200 Southpark Blvd, Suite 209, Saint Augustine, Florida
  - Hanger Clinic - 215 First Street North, Suite 300A, Winter Haven, Florida
  - Hanger Clinic - 607 N. Jefferson Street, Albany, Georgia
  - Hanger Clinic - 1050 Buford Rd, Ste 106, Cumming, Georgia
  - Hanger Clinic - 778 Riverside Drive, Macon, Georgia
  - Hanger Clinic - 1215A Merchant Way, Statesboro, Georgia
  - Hanger Clinic - 11346 S Cicero Ave, Alsip, Illinois
  - Hanger Clinic - 2835 N Sheffield Ave, Ste 301, Chicago, Illinois
  - Hanger Clinic - 1551 Bond Street, Suite 111, Naperville, Illinois
  - Hanger Clinic - 401 Harrison Street, Oak Park, Illinois
  - Hanger Clinic - 355 W Carpenter St., Springfield, Illinois
  - Hanger Clinic - 4821 Old National Road East, Suite A, Richmond, Indiana
  - Hanger Clinic - 4505 Utica Ridge Rd, Bettendorf, Iowa
  - Hanger Clinic - 866 5th Ave SE, Cedar Rapids, Iowa
  - Hanger Clinic - 330 Laurel St. #1300, Des Moines, Iowa
  - Hanger Clinic - 804 Kenyon Road, Fort Dodge, Iowa
  - Hanger Clinic - 645 East Crawford St, Salina, Kansas
  - Hanger Clinic - 410 N. Hillside, Suite 100, Wichita, Kansas
  - Hanger Clinic - 8522 Summa Ave, Baton Rouge, Louisiana
  - Hanger Clinic - 940 Kaliste Saloom, Lafayette, Louisiana
  - Hanger Clinic - 1010 Stillwater Ave, Ste 106, Bangor, Maine
  - Hanger Clinic - 959 Brighton Ave., Portland, Maine
  - Hanger Clinic - 1001 Cromwell Bridge Rd, Suite 108, Towson, Maryland
  - Hanger Clinic - 100 Erdman Way, STE 100, Leominster, Massachusetts
  - Hanger Clinic - 100 Milk Street, Suite 120, Methuen, Massachusetts
  - Hanger Clinic - 1985 Main Street, Springfield, Massachusetts
  - Hanger Clinic - 225 South Michigan Ave Suite B, Big Rapids, Michigan
  - Hanger Clinic - 1903 23rd Ave, Meridian, Mississippi
  - Hanger Clinic - 502 Council Circle, Tupelo, Mississippi
  - Hanger Clinic - 3065 William Street, Suite 205, Cape Girardeau, Missouri
  - Hanger Clinic - 150 St Peters Centre Blvd, City of Saint Peters, Missouri
  - Hanger Clinic - 2340 E. Meyer Blvd, Building 2, Suite 394, Kansas City, Missouri
  - Hanger Clinic - 65 Medical Park Drive, Suite 3, Helena, Montana
  - Hanger Clinic - 1001 S 70th St Ste 110, Lincoln, Nebraska
  - Hanger Clinic - 9109 Blondo Street, Omaha, Nebraska
  - Hanger Clinic - 17500 Burke St, Suite 100, Omaha, Nebraska
  - Hanger Clinic - 7250 Peak Drive, STE 120, Las Vegas, Nevada
  - Hanger Clinic - 961 Matley Ln Ste 100, Reno, Nevada
  - Hanger Clinic - New Hampshire - 7 Marsh Brook Dr Ste 201, Somersworth, New Hampshire
  - Hanger Clinic - 715 Dr Martin Luther King Jr Ave NE Ste, Albuquerque, New Mexico
  - Hanger Clinic - 1882 Winton Road South, Suite 6, Rochester, New York
  - Hanger Clinic - 5502 Brush Hollow Rd., Westbury, New York
  - Hanger Clinic - 2219 E. 7th St., Charlotte, North Carolina
  - Hanger Clinic - 1399 Westgate Center Dr, Winston-Salem, North Carolina
  - Hanger Clinic - One Elizabeth Place Suite 300, Dayton, Ohio
  - Hanger Clinic - 660 Wessel Drive, Fairfield, Ohio
  - Hanger Clinic - 6001 Landerhaven Dr Ste A, Mayfield Heights, Ohio
  - Hanger Clinic - 423 Normal St., East Stroudsburg, Pennsylvania
  - Hanger Clinic - 40 Berkshire Ct STE 2, Wyomissing, Pennsylvania
  - Hanger Clinic - 305 E Greenville St, Anderson, South Carolina
  - Hanger Clinic - 1739 Blanding St., Columbia, South Carolina
  - Hanger Clinic - 779 W. Forest Ave, Jackson, Tennessee
  - Hanger Clinic - 502 Princeton Rd, Johnson City, Tennessee
  - Hanger Clinic - 6300 Baum Dr, Knoxville, Tennessee
  - Hanger Clinic - 266 Cherokee Professional Park, Maryville, Tennessee
  - Hanger Clinic - 7 North Bellevue Blvd, Memphis, Tennessee
  - Hanger Clinic - 8000 State Highway 242, Suite 100, Conroe, Texas
  - Hanger Clinic - 3910 Gaston Ave STE 150, Dallas, Texas
  - Hanger Clinic - 320 West Water St, Suite D, Kerrville, Texas
  - Hanger Clinic - 4001 N Mays St. Ste 1200, Round Rock, Texas
  - Hanger Clinic - 1139 S.E. Military Dr., Suite 111, San Antonio, Texas
  - Hanger Clinic - 1400 College St, Ste 7, Sulphur Springs, Texas
  - Hanger Clinic - 17490 Hwy 3 Unit 100A, Webster, Texas
  - Hanger Clinic - 2785 East 3300 South, Salt Lake City, Utah
  - Hanger Clinic - 704 Thimble Shoals Blvd. Suite 400-B, Newport News, Virginia
  - Hanger Clinic - 5809 West Norfolk Road, Portsmouth, Virginia
  - Hanger Clinic - 1516 Hudson Street, Suite 105, Longview, Washington
  - Hanger Clinic - 401 SW 41st ST, Renton, Washington
  - Hanger Clinic - 4407 MacCorkle Ave SE, Charleston, West Virginia
  - Hanger Clinic - 5027 Green Bay Rd, Suite 124, Kenosha, Wisconsin
  - Hanger Clinic - 3440 Losey Blvd S, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No